CLINICAL TRIAL: NCT06932198
Title: Randomized, Single Oral Dose, Two-period, Two-treatment, Two-sequence Open-label, Crossover, Bioequivalence Study to Compare Selexipag 400mcg Film Coated Tablets (400 mcg Selexipag) Versus Uptravi® 400mcg Film Coated Tablets (400 mcg Selexipag), in Healthy Subjects Under Fed Conditions
Brief Title: Bioequivalence Study to Compare Selexipag 400mcg Film Coated Tablets (400 mcg Selexipag) Versus Uptravi® 400mcg Film Coated Tablets (400 mcg Selexipag)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1358-2024
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — selexipag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selexipag Film Coated Tablets (Experimental): Selexipag 400mcg Film Coated Tablets (400mcg Selexipag)
  Interventions: Drug: Selexipag Film Coated Tablets
- Uptravi® Film Coated Tablets (Active Comparator): Uptravi® 400mcg Film Coated Tablets (400mcg Selexipag)
  Interventions: Drug: Uptravi® Film Coated Tablets

INTERVENTIONS:
Drug: Selexipag Film Coated Tablets — 1 tablet
  Arms: Selexipag Film Coated Tablets
Drug: Uptravi® Film Coated Tablets — 1 tablet
  Arms: Uptravi® Film Coated Tablets

SUMMARY:
Randomized, single oral dose, two-period, two-treatment, two-sequence open-label, crossover, bioequivalence study to compare Selexipag 400mcg Film Coated Tablets (400 mcg Selexipag) versus Uptravi® 400mcg Film Coated Tablets (400 mcg Selexipag), in healthy subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* The subject is Caucasian & aged between eighteen to fifty (18-50), both inclusive.
* The subject is within the limits for his/her height & weight as defined by the body mass index range (18.5 - 30.0 Kg/m2).
* The subject is willing to undergo the necessary pre- & post- medical examinations set by this study.
* The results of medical history, physical examination, vital signs & conducted medical laboratory tests are normal as determined by the clinical investigator.
* The subject tested negative for Hepatitis B (HBsAg), Hepatitis C (HCVAb) and human immunodeficiency virus (HIVAb).
* There is no evidence of psychiatric disorder, antagonistic personality, and poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* The subject is able to understand and willing to sign the informed consent form.
* For female subjects: negative serum pregnancy test and the married woman is using two reliable contraception methods and should be non-lactating.
* The subject has normal cardiovascular system & normal ECG with normal QT interval corrected for heart rate according to Bazett's formula.
* The subject kidney and liver (AST & ALT enzymes) functions tests are within normal range. (Creatinine is accepted if below the reference range after being evaluated by the clinical investigator as clinically not significant).
* The subject Haematology test results are within normal range & RBC indices are within 5% of the normal range.
* The subject blood pressure is ≥ 110/70 mmHg before dosing.
* The subject has normal thyroid gland function.

Exclusion Criteria:

* The subject is a heavy smoker (more than 10 cigarettes per day).
* The subject has a history of or concurrent abuse of alcohol.
* The subject has a history of or concurrent abuse of illicit drugs.
* The subject has a history of hypersensitivity and/or contraindications to the study drug and any related compounds.
* The subject has suffered an acute illness one week before dosing.
* The subject has been hospitalized within three months before the study or during the study.
* The subject is on special diet (for example subject is vegetarian.)
* The subject has consumed caffeine or xanthine containing beverages or foodstuffs within two days before dosing and until 72 hours after dosing in both study periods.
* The subject has taken a prescription medication within two weeks or even an over the counter product (OTC) within one week before dosing in each study period and any time during the study, unless otherwise judged acceptable by the clinical investigator.
* The subject has taken grapefruit/orange containing beverages or foodstuffs within seven (7) days before first dosing and any time during the study.
* The subject has been participating in any clinical study (e.g. pharmacokinetics, bioavailability and bioequivalence studies) within the last 80 days prior to the present study.
* The subject has donated blood within 80 days before first dosing.
* The subject has a history or presence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinal, immunological, dermatological, neurological, musculoskeletal, ocular or psychiatric diseases.
* The subject has consumed drugs that may affect pharmacological or pharmacokinetic properties of Selexipag (for example: gemfibrozil, clopidogrel, deferasirox, teriflunomide, rifampicin, carbamazepine, phenytoin, valproic acid, probenecid, fluconazole, lopinavir/ritonavir). two weeks before dosing, during the study and two weeks after dosing.
* The subject has recently experienced significant blood loss or fluid loss such as severe diarrhoea or vomiting.

Note: Subjects, who were screened for another study and were not enrolled, might be recruited for this study provided they meet the acceptance criteria of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | 72 hours
  two-sided 90 % CI for the test to reference ratio of the population means is within 80.00 - 125.00 % for each of the Ln-transformed data Cmax
AUC from time 0 to last collection time t (AUC0 - t) | 72 hours
  two-sided 90 % CI for the test to reference ratio of the population means is within 80.00 - 125.00 % for each of the Ln-transformed data AUC0-t

SECONDARY OUTCOMES:
Time to reach maximum concentration Cmax (Tmax) | 72 hours
  Descriptive Statistics
half-life (Thalf) | 72 hours
  Descriptive Statistics

CONTACTS AND LOCATIONS:
Locations (1):
- ACDIMA Center, Amman, Jordan